CLINICAL TRIAL: NCT04097756
Title: A Phase I Study of LX-039 Tablets in Postmenopausal Patients With ER+, HER2- Advanced Breast Cancer After Failure of Endocrine Therapy
Brief Title: A Phase I Study of LX-039 Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Luoxin Pharmaceutical Group Stock Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OE861801
Record Dates: First submitted 2019-07-29; First posted 2019-09-20 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2020-10

CONDITIONS: Advanced Breast Cancer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part1：dose escalation (Experimental): The investigational product for this study is LX-039 tablets,which can be administered orally. 6~8 ascending dose level until MTD and the specification included 50 mg, 100 mg, 200 mg, 400 mg, 600 mg , 800 mg,1050 mg and 1400 mg. LX-039 tablets will be administered in a therapeutic cycle of 28 days once a day orally. The subjects will continue therapy with LX-039 if good safety and tolerability were assessed by investigators after one cycle treatment. The treatment will continue until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
  Interventions: Drug: LX-039 tablets
- Part 2：dose expansion (Experimental): 2~3 selected tolerable dose will be selected according to the tolerance and FES PET results of dose escalation phase.The subjects will continue therapy with LX-039 if good safety and tolerability were assessed by investigators after one cycle treatment. The treatment will continue until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
  Interventions: Drug: LX-039 tablets

INTERVENTIONS:
Drug: LX-039 tablets — orally once daily until disease progression, unacceptable toxicity, withdrawal of consent, or study termination

SUMMARY:
This is a phase I dose escalation and expansion study in patients with ER+, HER2- advanced breast cancer to explore the tolerance, PK/PD(pharmacokinetics/pharmacodynamics) profiles and preliminary anti-tumor activity of different doses of LX-039 tablets. The trial consists of two parts, dose escalation and dose expansion. Part 1 is the dose escalation phase with initial 6 dose groups, and "3 + 3" design is used to explore MTD of the drug; Part 2 is the dose expansion phase with 2 ~ 3 doses selected for expansion according to the escalation results of Part 1, and more subjects are enrolled to further observe the tolerance and preliminary anti-tumor activity of the drug. After the completion of dose expansion, the recommended phase II dose (RP2D) will be determined after discussion based on the obtained tolerance and PK/PD data.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to read and sign the informed consent form.
2. Adult females (aged ≥18 and ≤75 years).
3. Be diagnosed with breast cancer confirmed by pathological examination.
4. Be histologically or cytologically confirmed estrogen receptor positive (ER+≥1% positive staining).
5. Be postmenopausal.
6. Subjects who have previously received endocrine therapy and obtained benefit.
7. ECOG(Eastern Cooperative Oncology Group) score ≤ 1.
8. Subjects in part2 of the study need to have measurable lesions that meet RECIST 1.1 criteria.
9. Has recovered from toxicity or injury from prior chemotherapy/radiotherapy .
10. Enough hematology and organ function.
11. Expected survival>3 months.

Exclusion Criteria:

1. Subjects with HER2-overexpressing breast cancer.
2. Subjects with known brain metastases or other central nervous system metastases that are symptomatic or untreated.
3. Patients with symptomatic advanced disease who have spread to the viscera and are at risk of life-threatening complications.
4. Subjects who received second-line or above chemotherapy.
5. Subjects with known allergy to this product or any of its components.
6. Subjects who previously used other estrogen receptor down regulators than fulvestrant.
7. Subjects who received endocrine therapy or other anti-tumor agent or radiotherapy within 4 weeks prior to study entry.
8. Subjects who received cell therapy or tumor vaccine therapy;
9. Subjects with severe immunosuppression .
10. Severe or uncontrolled disease.
11. Subjects with diseases or abnormalities that may affect the administration and absorption of drugs.
12. Subjects with other malignancy within 5 years prior to study entry.
13. Subjects with other high risks of thrombosis or require long-term use of antiplatelet drugs.
14. Subjects with history of definite neurological or psychiatric disorders in the past.
15. Subjects who are HIV(human immunodeficiency virus) antibody positive, HBsAg(hepatitis B surface antigen) positive or HCV(hepatitis C virus)antibody positive.
16. Subjects with other uncontrolled malignant/non-malignant diseases, significant laboratory abnormalities, participation in the study may increase the risk.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
To explore the tolerance of LX-039 in ER +, HER2 - patients with advanced breast cancer | DLT observation period(5 weeks for dose escalation, 4 weeks for dose expansion)
  Incidence of dose limiting toxicities (DLTs)

SECONDARY OUTCOMES:
The safety of LX-039 in ER +, HER2 - patients with advanced breast cancer | through study completion,an average of 1 year
  Number of participants with treatment related. adverse events as assessed by CTCAE v5.0
To explore the efficacy of LX-039 in ER +, HER2 - patients with advanced breast cancer according to Recist 1.1. | through study completion，an average of 1 year.
  Objective response rate (ORR)
To explore the efficacy of LX-039 in ER +, HER2 - patients with advanced breast cancer according to Recist 1.1. | through study completion，an average of 1 year.
  proportion of subjects with complete response (CR）
To explore the efficacy of LX-039 in ER +, HER2 - patients with advanced breast cancer according to Recist 1.1. | through study completion，an average of 1 year.
  proportion of subjects with partial response (PR）
To explore the efficacy of LX-039 in ER +, HER2 - patients with advanced breast cancer according to Recist 1.1. | through study completion，an average of 1 year.
  proportion of subjects with stable disease (SD)
To explore the efficacy of LX-039 in ER +, HER2 - patients with advanced breast cancer according to Recist 1.1. | through study completion，an average of 1 year.
  proportion of subjects with progressive disease (PD)
To explore the efficacy of LX-039 in ER +, HER2 - patients with advanced breast cancer according to Recist 1.1. | through study completion，an average of 1 year.
  duration of response (DoR)
To explore the efficacy of LX-039 in ER +, HER2 - patients with advanced breast cancer according to Recist 1.1. | through study completion，an average of 1 year.
  disease control rate (DCR)
To explore the efficacy of LX-039 in ER +, HER2 - patients with advanced breast cancer according to Recist 1.1. | through study completion，an average of 1 year.
  clinical benefit rate (CBR)
To explore the efficacy of LX-039 in ER +, HER2 - patients with advanced breast cancer according to Recist 1.1. | through study completion，an average of 1 year.
  time to progression (TTP)
To explore the efficacy of LX-039 in ER +, HER2 - patients with advanced breast cancer according to Recist 1.1. | through study completion，an average of 1 year.
  progression-free survival (PFS)
To explore the efficacy of LX-039 in ER +, HER2 - patients with advanced breast cancer according to Recist 1.1. | through study completion，an average of 1 year.
  overall survival (OS)
Comparison of changes in maximum uptake ability of FES(progression free survival) in breast cancer lesions before and after treatment with LX-039 by PET(positron emission tomography) scan (performed in some subjects) | Up to the third day of Cycle 2(each cycle is 28 days)
  Decrease in SUVmax in comparison with that before treatment
PK profiles after a single dose of LX-039 | Up to the third day of Cycle 0(Cycle 0 is 7 days)
  Peak Concentration (Cmax)
PK profiles after a single dose of LX-039 | Up to the third day of Cycle 0(Cycle 0 is 7 days)
  Peak Time (Tmax)
PK profiles after a single dose of LX-039 | Up to the third day of Cycle 0(Cycle 0 is 7 days)
  Elimination Half-life (t1/2)
PK profiles after a single dose of LX-039 | Up to the third day of Cycle 0(Cycle 0 is 7 days)
  Eliminate Rate Constant (Kel)
PK profiles after a single dose of LX-039 | Up to the third day of Cycle 0(Cycle 0 is 7 days)
  Mean Residence Time (MRT)
PK profiles after a single dose of LX-039 | Up to the third day of Cycle 0(Cycle 0 is 7 days)
  Area under plasma Concentration-time curve from 0 time to 24 hours (AUC0-24h)
PK profiles after a single dose of LX-039 | Up to the third day of Cycle 0(Cycle 0 is 7 days)
  Area under plasma Concentration-time curve from 0 time to sampling time t of the last measurable concentration (AUC0-last)
PK profiles after a single dose of LX-039 | Up to the third day of Cycle 0(Cycle 0 is 7 days)
  Area under plasma Concentration-time curve from administration (0) to infinity (AUC0-inf)
PK profiles after a single dose of LX-039 | Up to the third day of Cycle 0(Cycle 0 is 7 days)
  Apparent Total Clearance (CL/F)
PK profiles after a single dose of LX-039 | Up to the third day of Cycle 0(Cycle 0 is 7 days)
  Apparent Volume of Distribution (Vd/F)
PK profiles after continuous administration of LX-039 | Up to the Second day of Cycle 2(each cycle is 28 days)
  Trough Concentration at Steady State (Css, min)
PK profiles after continuous administration of LX-039 | Up to the Second day of Cycle 2(each cycle is 28 days)
  Peak Concentration at Steady State (Css, max)
PK profiles after continuous administration of LX-039 | Up to the Second day of Cycle 2(each cycle is 28 days)
  Average Concentration at Steady State (Css, av)
PK profiles after continuous administration of LX-039 | Up to the Second day of Cycle 2(each cycle is 28 days)
  Peak Time (Tss, max)
PK profiles after continuous administration of LX-039 | Up to the Second day of Cycle 2(each cycle is 28 days)
  Apparent Volume of Distribution at steady state (Vss/F)
PK profiles after continuous administration of LX-039 | Up to the Second day of Cycle 2(each cycle is 28 days)
  Steady-state Clearance Half-life (tss,1/2)
PK profiles after continuous administration of LX-039 | Up to the Second day of Cycle 2(each cycle is 28 days)
  Total Body Clearance (CLss/F)
PK profiles after continuous administration of LX-039 | Up to the Second day of Cycle 2(each cycle is 28 days)
  Coefficient of Fluctuation (DF)
PK profiles after continuous administration of LX-039 | Up to the Second day of Cycle 2(each cycle is 28 days)
  Area under Plasma Concentration-time Curve at Steady State (AUCss)
PK profiles after continuous administration of LX-039 | Up to the Second day of Cycle 2(each cycle is 28 days)
  Accumulation Coefficient (Rac)

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Lu J, Chan CC, Sun D, Hu G, He H, Li J, Dong J, Liu K, Shen L, Hu L, Gu Q, Chen S, Wang T, Gong T, Tang W, Li X, Zhu X, Zeng X, Zhu Y, Xia Y, Huang Y, Zhu Y, Liu Z, Ding CZ. Discovery and preclinical profile of LX-039, a novel indole-based oral selective estrogen receptor degrader (SERD). Bioorg Med Chem Lett. 2022 Jun 15;66:128734. doi: 10.1016/j.bmcl.2022.128734. Epub 2022 Apr 15. PMID 35436589